CLINICAL TRIAL: NCT00161525
Title: Perfluorocarbon Gases for the Repair of Retinal Detachments.
Brief Title: Pneumatic Displacement of Subretinal Hemorrhage With Perfluorocarbon Gases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The Edward Grayson Fund for Retinal Research (Unknown)
Responsible Party: Harvey A. Lincoff M.D., Weill Cornell Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1095-053
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Subretinal Hemorrhage and Exudative Maculopathy
Keywords: Subretinal Hemorrhage, Perfluorocarbon gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pneumatic displacement — Pneumatic displacement of the subretinal hemorrhages is attempted with an intravitreous injection of 0.4 ml of pure C2F6 or 2 injections of 0.2 ml on subsequent days. The gas is withdrawn from a laboratory cylinder through a millipore filter and injected into the eye through a 30 gauge needle inserted 4.0 mm posterior to the limbus in the superior temporal quadrant. The tip of the needle is monitored in the vitreous by indirect ophthalmology prior to injecting the gas.Post injections the central retinal artery is examined whether is patent.The intraocular gas expands 3.3 times over the next 3 days to create a 40% bubble.The patient is asked to assume a gaze position 40° below the horizontal for 20 minutes every hour while awake and to sleep on 2 pillows with his head turned to the right.

SUMMARY:
Subretinal hemorrhage in the macula causes a significant loss of vision. This hemorrhage can be displaced by the use of a small volume of pure perfluorocarbon gas injected into the vitreous, which expands to a 40% gas bubble in the eye. When the patient gazes 40 to 60 degree below the horizontal, the gas bubble covers the hemorrhage and gravity displaces it rapidly. This position of gaze is easier for the patient than the face down position traditionally recommended.A vector of gravity force tangential to the sclera brings about this displacement. The procedure can improve vision quickly, reduce unwanted degenerative changes in the macula because of the persistent macular hemorrhage and improves the chances of treating of the underlying cause for the subretinal hemorrhage by laser or other means.

DETAILED DESCRIPTION:
This protocol was designed to determine the optimum position of the gaze for pneumatic displacement of subretinal hemorrhage (SRH) in the macula. A geometrical analysis of the forces that act upon a SRH in the presence of an intraocular gas bubble was analyzed and it was concluded that the displacement was due to the effect of gravity on the SRH immersed in gas. This was followed by a prospective trial of positions of gaze and volumes of gas calculated to be optimum for displacement. The eyes of consecutive patients with SRH in the macula will had an intravitreal injection of pure perfluorocarbon gas sufficient to provide a 40% bubble after expansion. The patients are instructed to gaze down 40° or 60° below the horizontal depending on the volume of gas for 20 minutes every hour. The SRH is displaced rapidly in the first week. Visual acuity usually improves but recovery can be limited by the presence of sub pigment epithelial hemorrhage, exudate or proliferation. A vector of the gravity force tangential to the sclera is the largest force acting to displace a subretinal hemorrhage within a gas bubble. 79% of the vertical gravity component is obtained at gaze 40° below the horizontal and requires volumes of intraocular gas not requiring prior removal of vitreous. Face down positioning in common practice has been an error and succeeds only if the patient has been non compliant.

5- STATUS

ELIGIBILITY:
Inclusion Criteria:

* Diminished vision secondary to subretinal hemorrhage in the macula or exudative maculopathy.

Exclusion Criteria:

* Patient unable to maintain gaze position for 20 minutes every waking hour for 7 days.
* Patient unable to sleep on their side or with head elevated 40 degrees.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2003-10; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Displacement of Subretinal Hemorrhage | 7 days after gas injection

SECONDARY OUTCOMES:
Improvement in visual acuity | 7 days after gas injection

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Lincoff, MD, Principal Investigator — New York Presbyterian Hospital, New York, NY 10021, United States
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Background] Johnson MW. Pneumatic displacement of submacular hemorrhage. Curr Opin Ophthalmol. 2000 Jun;11(3):201-6. doi: 10.1097/00055735-200006000-00009. PMID 10977228